CLINICAL TRIAL: NCT02223585
Title: Gut Microbial Response to Well-balanced Diet With Emphasis on Animal or Vegan Protein
Brief Title: Gut Microbiota and Proteins Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13.28.MET
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Gut microbial; response; to protein-based; diet; challenges; population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cross-over single arm (Experimental)
  Interventions: Other: Animal-based protein diet; Other: Vegan-based protein diet

INTERVENTIONS:
Other: Animal-based protein diet
Other: Vegan-based protein diet

SUMMARY:
Gut microbiota are involved in the regulation of mammalian metabolic pathways through host-microbiota metabolic, signaling, and immune-inflammatory interactions that physiologically connect the gut, liver, brain, and other organs. Correlation of these metabotypes with gut microbial profiles facilitates deciphering inherent host-microbe relationships.

Microbiome sequencing have generated novel insights into the role of gut microbial composition in health and disease, but are limited in addressing the microbial contribution to host metabolism and the gut microbial dysbiosis in disease.

This is an exploratory trial, aiming to examine how gut microbial conditions determine response to dietary challenge by measuring urine, plasma and stool metabolites resulting from metabolism of protein, polyamines and bile acids in combination with stool bacterial composition. The focus of this trial is to evaluate impact of protein based food challenges, based on cross-over design of two diet challenges of animal and vegan protein sources.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Regular bowl movement (at least once every 1-2 days)
* Between 18 and 55 years old
* BMI between 18.5 and 27 kg/m2 (inclusive)
* Willing and able to sign written informed consent prior to trial entry

Exclusion Criteria:

* Clinically relevant digestive, renal or metabolic disease, as determined by the medical (screening) visit and a standard blood chemistry analysis (glucose, total cholesterol, LDL, HDL, triglycerides, Aspartate aminotransferase (ASAT), Alanine aminotransferase (ALAT), gamma glutamyl transferase (Gamma-GT), C reactive protein (CRP), creatinine)
* Undergoing regular medical treatment, pain-killers accepted, based on the medical questionnaire
* Special diets: vegetarian, high protein or weight loss program (anamnesis)
* Pregnancy (anamnesis)
* Food allergy
* Participation in a cholesterol management program with functional foods like food supplement enriched in omega-3 fatty acids, dairy products enriched with phytosterols (margarines, yoghurts), evaluated during the medical visit
* Practicing more than 5 moderated physical activity per week
* Smoker (anamnesis)
* Have a high alcohol consumption (more than 2 drinks/day) (anamnesis)
* Consumption of illicit drugs, (anamnesis)
* Having given blood within the last month, or willing to make a blood donation until one month following the end of the study
* Subject who cannot be expected to comply with the study procedures, including consuming the test products.
* Currently participating or having participated in another clinical trial during the last month prior to the beginning of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Intra-individual plasma, stools, and urine omics to acute controlled feeding | 3-Day baseline, 3-Day diet challenge 1, 1-Day baseline after challenge 1 washout, 3-Day diet challenge 2, 1-Day baseline after challenge 2 washout
  Metabonomics on fasting blood, urine, and stools and microbiota composition by 1. defining individual baseline (3-Day baseline before start of diet challenges); 2. Examining effect of the dietary challenges (3-Day diet challenge vs. Baseline); 3. Examining global dietary effect (baseline after challenge 2 vs. baseline after challenge 1) and stability of dietary effect (3rd day of each diet challenge vs. baseline after the challenge)
Intra-individual plasma biochemistry response to acute controlled feeding | Day 1 and 3 of diet challenge 1, 1-Day baseline after challenge 1 washout, Day 1 and 3 of diet challenge 2, 1-Day baseline after challenge 2 washout
  To evaluate effect of the dietary challenges (Day 3 vs Day1 of each diet challenge), the global dietary effect (baseline after challenge 2 vs. the baseline after challenge 1, Day 1 of diet challenge 1), stability of the dietary effect (3rd day of each diet challenge vs. baseline after the challenge)

SECONDARY OUTCOMES:
Subject's omics adaptation phase to a controlled diet Subject's omics adaptation phase to a controlled diet | 3-Day diet challenge 1 and 2
  Through analysis of metabonomics on fasting blood, daytime blood, urine, and stools and microbiota composition
Comparison of intra-individual daytime plasma response amongst diets and free living restricted diets | 3-Day baseline before start of diet challenges, 3-Day diet challenge 1, 1-Day baseline after challenge 1 washout, 3-Day diet challenge 2, 1-Day baseline after challenge 2 washout
  Through analysis of metabonomics on fasting blood, daytime blood, urine, and stools and microbiota composition
Pairing of gut microbial metabolite to gut microbial composition to generate concept on gut functional system to be followed-up in future studies | 3-Day baseline before start of diet challenges, 3-Day diet challenge 1, 1-Day baseline after challenge 1 washout, 3-Day diet challenge 2, 1-Day baseline after challenge 2 washout
  Through analysis of metabonomics on fasting blood, daytime blood, urine, and stools and microbiota composition
Pairing dietary intake and preferences with subjects response in Omics endpoints | 3-Day baseline before start of diet challenges, 3-Day diet challenge 1, 1-Day baseline after challenge 1 washout, 3-Day diet challenge 2, 1-Day baseline after challenge 2 washout
  Through analysis of metabonomics on fasting blood, daytime blood, urine, and stools and microbiota composition and 3- Days dietary recall during diet challenges and food frequency questionnaire at baseline before start of diet challenges

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, PhD, PD Dr, Principal Investigator — Metabolic Unit, Clinical Development Unit, Nestec
Locations (1):
- Metabolic Unit, Clinical Development Unit, Nestec, Lausanne, Switzerland

REFERENCES:
- [Derived] Draper CF, Tini G, Vassallo I, Godin JP, Su M, Jia W, Beaumont M, Moco S, Martin FP. Vegan and Animal Meal Composition and Timing Influence Glucose and Lipid Related Postprandial Metabolic Profiles. Mol Nutr Food Res. 2019 Mar;63(5):e1800568. doi: 10.1002/mnfr.201800568. Epub 2019 Feb 21. PMID 30724465